CLINICAL TRIAL: NCT06432946
Title: Effect of Two Facilitating Interventions on the Acceptability and Usability Towards a Sensing-glove System to Measure Force-time Characteristics of Spinal Manipulative Therapy: a Mixed-methods Cross-over Study
Brief Title: Sensing-glove System in Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Isabelle Pagé, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UQTR_IP_Acceptabilite_2021
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Spinal Manipulation
Keywords: Chiropractic; Manual therapy; Acceptability; Usability; Force-time characteristics
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Participants will undergo two interventions consecutively, with the order of evaluation randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video followed by practice (Experimental): Participants will initially view a 7-minute informational video followed by a 20-minute supervised practice session with the sensing-glove system. Acceptability and usability perception will be assessed after each intervention.
  Interventions: Other: Video; Other: Practice session
- Practice followed by video (Experimental): Participants will initially participate in a 20-minute supervised practice session with the sensing-glove system followed by viewing a 7-minute informational video. Acceptability and usability perception will be assessed after each intervention.
  Interventions: Other: Video; Other: Practice session

INTERVENTIONS:
Other: Video — A 7-minute video demonstrating the sensing-glove system, how it can be used to assess manual therapy biomechanics, and its relevance in research and clinical contexts. The video was created by the research team via a voiceover PowerPoint presentation.
Other: Practice session — A 20-minute practice session during which participants received verbal information about the sensing-glove system. While wearing the sensing glove, participants performed palpation and manual therapy techniques (palpation, spinal mobilization/manipulation to the cervical and thoracic spine) on a human-sized manikin, guided by the researcher.

SUMMARY:
The objective of this clinical trial is to assess manual therapists' attitudes towards using a sensing-glove system for measuring spinal manipulation force and to compare the effectiveness of two interventions in enhancing their attitudes. The primary questions it aims to address are:

* Are manual therapists receptive to employing a sensing-glove system to measure the force applied during spinal manipulations on patients?
* Can we enhance manual therapists' attitudes towards this system through either a brief informational video demonstration or a supervised practice session with the system?

Researchers will compare the impact of a 7-minute informational video to that of a 20-minute supervised practice session to determine if manual therapists' attitudes towards the use of a sensing-glove while treating their patients can be positively influenced.

Participants will:

* Engage in a single experimental session.
* Complete a questionnaire at the beginning of the experimental session.
* Undergo one of the two interventions and promptly complete two questionnaires following this intervention.
* Undergo the other intervention and promptly complete the same two questionnaires following this intervention.

DETAILED DESCRIPTION:
This study aimed to evaluate manual therapists' acceptability of a sensing-glove system for measuring spinal manipulation's force-time characteristics and compare the effectiveness of two interventions in enhancing their acceptability and usability perception. Participants will undergo two acceptability-enhancing interventions in randomized order: a 7-minute informational video and a 20-minute supervised practice session. At the start of the session and after each intervention, the acceptability and perception of usability towards the system will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed chiropractor or a last-year intern in a University outpatient chiropractic clinic

Exclusion Criteria:

* Reported any upper limb injury preventing them from executing manual therapies during the time of the study
* Previous experience with the sensing-glove system

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | Immediately following each intervention and at baseline
  French version of the questionnaire based on the extended version of the Unified Theory of Acceptance and Use of Technology (UTAUT2). A higher score indicates a higher level of acceptability.
Usability | Immediately following each intervention
  French version of the System usability scale (F-SUS). A higher score indicates a higher level of usability.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No